CLINICAL TRIAL: NCT02716545
Title: the Efficiency of Endoscopic Treatment for Recurrent Small Intestinal Bleeding Due to Gastrointestinal Vascular Malformation: the Study of the Bleeding Risks Stratification Model and Endoscopic Treatment
Brief Title: the Efficiency of Endoscopic Treatment for Recurrent Small Intestinal Bleeding Due to Gastrointestinal Vascular Malformation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhizheng Ge, Director of digestive endoscopy centre of Renji hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rj(2015)088K-b
Record Dates: First submitted 2016-03-11; First posted 2016-03-23 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Gastrointestinal Vascular Malformation
Keywords: Gastrointestinal vascular malformation; Endoscopic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endoscopic Intervention Group (Experimental): Endoscopic therapy
  Interventions: Device: balloon assisted enteroscopy

INTERVENTIONS:
Device: balloon assisted enteroscopy — Patients with recurrent bleeding (>2 times for one year) will undergo balloon assisted enteroscopy and be treated with endoscopic therapy if necessary. Currently available endoscopic modalities are argon laser, bipolar electrocoagulation (BiCAP), band ligation, cryotherapy, radiofrequency ablation and argon plasma coagulation (APC). Among these options, APC is the most promising.

SUMMARY:
Gastrointestinal vascular malformation (GIVM), which is an important cause of acute or chronic gastrointestinal bleeding, consequently is in dire of effective treatment. The investigators' previous study first confirmed thalidomide treatment of GIVM bleeding was safe and effective. This trial intends to investigate the efficiency of endoscopic intervention to the hemorrhage due to GIVM. What more, the research tends to suggest standardizing clinical paths for small bowel bleeding due to GIVM.

DETAILED DESCRIPTION:
This multi-institutional clinical trial investigates the efficacy of endoscopic intervention to the recurrent small intestinal hemorrhage due to GIVM. Patients with recurrent bleeding (>2 times for one year) will undergo balloon assisted enteroscopy and be treated with endoscopic therapy if necessary. The hierarchical primary endpoints were the difference in yearly Bleeding times, followed (if significant) by the difference in Blood Transfusions, Total Transfused Red Cell Requirements, yearly bleeding Episodes, Bleeding Duration, yearly average Hemoglobin (Hb) level, hospitalization and iron requirement. The study will be done at 10 centers in China.

ELIGIBILITY:
Inclusion Criteria:

The patients should sign informed consent and be informed of the specific trial plan;

* The patients should have the China nationality;
* The patients should be aged from 18 to 70 years old, male or female;
* The intestinal vascular lesions should be found by capsule endoscopy, and / or balloon assisted enteroscopy; OR the patients should present with persistent and recurrent bleeding, while the bleeding lesions are unable to be located by all these examinations mention above;
* The patients should present with persistent and recurrent bleeding (>=2 times for one year);
* Hb levels should decreased 10% lower than baseline.
* The patient is willing to comply with the instructions and have the ability to complete the study of research program.

Exclusion Criteria:

patients associated with varicosity due to cirrhosis of the liver; Or patients with uncontrolled hypertension, hyperglycemia, or other severe diseases;

* patients with a history of severe peripheral neuropathy, seizures, rheumatoid immune disease, or thromboembolic disease;
* patients with indications which should constantly use non-steroidal anti-inflammatory drugs, anticoagulants and anti-platelet or acetyl salicylic acid preparation, ginkgo, Echinacea, Chinese herbal medicine composition, other anti-angiogenesis drugs;
* patients with malignant or severe heart disease (uncontrolled angina and/or myocardial infarction, congestive heart failure within 3 months before recruiting, etc.), lung disease (respiratory failure), kidney, pancreatic, liver disease or other diseases that researchers evaluated as affect the judgment of the treatment;
* previously small intestinal bowel resection surgery;
* serious life-threatening gastrointestinal bleeding requiring immediate surgical treatment;
* alcohol and/or drug abuse, addiction or rely on) or the doctor determine compliance claim;
* patients had been recruited into other clinical research within 6 months;
* personnel related to this study;
* patients have no legal behavior ability or self-knowledge; Or patients refuse into groups.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Participants Whose yearly Rebleeding times Decreased From Baseline by ≥ 50% | up to 3 yrs

SECONDARY OUTCOMES:
Difference of patients completely cured | up to 3 yrs
  The cessation of bleeding was defined as repeated negative fecal occult blood test (FOBT) (monoclonal colloidal gold color technology) during our observation period. Rebleeding was defined based on a positive FOBT at any visit after treatment
difference in Blood Transfusions Requirements | up to 3 yrs
difference in Total Transfused Red Cell Requirements | up to 3 yrs
difference in yearly bleeding Episodes | up to 3 yrs
difference in yearly mean Hemoglobin (Hb) level | up to 3 yrs
numbers of patients requiring hospitalization | up to 3 yrs
difference of yearly hospitalization times | up to 3 yrs
difference of the number of days in hospital yearly | up to 3 yrs
difference in mean iron requirements | up to 3 yrs

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Renji Hospital, Shanghai Institute of Digestive Diseases, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No